CLINICAL TRIAL: NCT03415295
Title: Association Between Trimethylamine-N-oxide Levels and Risk of Gestational Diabetes Mellitus
Brief Title: Association Between Trimethylamine-N-oxide and Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Director, Huazhong University of Science and Technology
Other Study IDs: SZSM201511007
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Gestational Diabetes
Keywords: Trimethylamine-N-oxide; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Maternal fasting blood samples were collected in anticoagulative tubes and centrifuged at 3000 rpm for 5 min. Then, the plasma was separated and stored at -80°C for subsequent analysis of TMAO and other blood parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: Gestational diabetes mellitus (GDM) was diagnosed according to the American Diabetes Association criteria, which is based on the "one-step" approach recommended by the International Association of Diabetes and Pregnancy Study Groups. All women underwent a 75g OGTT in the morning after an overnight fast, with plasma glucose measurement fasting and at 1 and 2 hours. The criteria for GDM diagnosis was to have at least one abnormal value: Fasting glucose ≥ 5.1 mmol/L (92 mg/dL), 1 h glucose ≥ 10.0 mmol/L (180 mg/dL), 2 h glucose ≥ 8.5 mmol/L (153 mg/dL).
  Interventions: Other: Plasma TMAO concentration
- Healthy pregnant control: Pregnant women with fasting glucose < 5.1 mmol/L (92 mg/dL), 1 h glucose < 10.0 mmol/L (180 mg/dL) and 2 h glucose < 8.5 mmol/L (153 mg/dL) were considered as healthy controls.
  Interventions: Other: Plasma TMAO concentration

INTERVENTIONS:
Other: Plasma TMAO concentration — Plasma TMAO concentrations were determined by stable isotope dilution liquid chromatography with online electrospray ionization tandem mass spectrometry on an AB SCIEX 4500 triple quadrupole mass spectrometer

SUMMARY:
Background: The microbiota-dependent metabolite trimethylamine-N-oxide (TMAO) has been reported as a novel and independent risk factor for the development of cardiovascular and metabolic diseases, but the association with gestational diabetes mellitus (GDM) remains unclear.

Objective: To investigate the association between plasma TMAO concentration and GDM in a two-phase study.

Design: The initial discovery phase included 866 pregnant women (433 GDM cases and 433 matched controls) in Wuhan China. Study participants were recruited from pregnant women who attended the outpatient clinics of the Department of Endocrinology, Tongji Hospital, to screen for GDM between August 2012 and April 2015, or pregnant women who visited the Hubei Maternal and Child Health Hospital or the Central Hospital of Wuhan for a routine antenatal checkup from May 2014 to November 2016. The inclusion criteria of participants were: age ≥ 20 years, gestational age between 24 and 32 weeks, no history of a diagnosis of diabetes or gestational diabetes, and no history of receiving pharmacological treatment known to affect glucose metabolism. An independent replication phase study was nested within an ongoing prospective cohort study, namely the Tongji Maternal and Child Health Cohort (TMCHC). Beginning in January 2013, women receiving prenatal care prior to 16 weeks of gestation were invited to join the TMCHC. Exclusion criteria included pre-pregnancy diabetes, clinically significant neurological, endocrinological or other systemic diseases and multiple pregnancies. All enrolled pregnant women received a regular prenatal checkup in hospital and underwent an oral glucose tolerance test (OGTT) during 24-32 weeks of gestation to screen for GDM. 276 members who developed GDM before May 2016 and had fasting blood collected before 20 weeks'gestation were included as cases in this analysis. Two controls were individually matched to each case from among women without GDM. These two studies were approved by the ethics committee of Tongji Medical College. All the participants gave informed written consent before they were included in the study. Plasma TMAO concentrations were determined by stable isotope dilution liquid chromatography with online electrospray ionization tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years;
* Screened for GDM during 24-32 weeks of gestation;
* With fasting blood samples collected before 20 weeks of gestation (only for nested case-control subjects).

Exclusion Criteria:

* History of a diagnosis of diabetes or gestational diabetes;
* History of receiving pharmacological treatment known to affect glucose metabolism;
* Clinically significant neurological, endocrinological or other systemic diseases and multiple pregnancies.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants enrolled were Chinese women. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation
Sampling Method: Probability Sample
Enrollment: 1694 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | During 24-32 weeks of gestation
  Glucose intolerance with onset or first diagnosis during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, Study Director — Department of Nutrition and Food Hygiene, School of Public Health, Huazhong University of Science and Technology

REFERENCES:
- [Derived] Li P, Zhong C, Li S, Sun T, Huang H, Chen X, Zhu Y, Hu X, Peng X, Zhang X, Bao W, Shan Z, Cheng J, Hu FB, Yang N, Liu L. Plasma concentration of trimethylamine-N-oxide and risk of gestational diabetes mellitus. Am J Clin Nutr. 2018 Sep 1;108(3):603-610. doi: 10.1093/ajcn/nqy116. PMID 30535087